CLINICAL TRIAL: NCT04519450
Title: Ultrasound Measurements of Accessory Respiratory Muscles in the Intensive Care Unit
Brief Title: Ultrasound of Accessory Respiratory Muscles
Status: Completed | Type: Observational
Sponsor: Osijek University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: OsijekUH-8
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2020-08

CONDITIONS: Mechanical Ventilation; Duration of Treatment; Survival
Keywords: Respiratory Muscles; Critical Care; Ultrasonography; Critical Care Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU patients without an with chronic respiratory diseases: The group will consist of >50 patients admitted to the intensive care unit, of which at least 20 with chronic respiratory diseases. Patients of both sexes, patients with and without chronic respiratory diseases, and also patients requiring mechanical ventilation were included and their demographic characteristics and outcomes registered. All patients will sign an informed consent form before inclusion in the prospective observational study.
  Interventions: Device: Mindray TE7 ultrasound machine

INTERVENTIONS:
Device: Mindray TE7 ultrasound machine — The study was performed using a Mindray TE7 ultrasound machine with the depth of the linear probe at 70 mm and gain of 90 dB; settings remained unchanged during the study. Measurements of the right m. sternocleidomastoideus, the right m. trapezius, and the right upper leg were taken, with the final value being the average of three measurements for each. The probe was set at the musculoskeletal ultrasound setting.
  Other Names: Mindray TE7

SUMMARY:
The aim of this study is to compare the diameter of accessory respiratory muscles in patients with respiratory diseases and patients without such diseases, and to determine whether there is a connection between the ultrasound-measured thickness of accessory respiratory muscles and time of mechanical ventilation, as well as whether there is a the connection between the measured thickness and the treatment outcome of patients in the Intensive Care Unit (ICU).

DETAILED DESCRIPTION:
An informed consent for the study was obtained from Ethics Committee, Osijek University Hospital, and Medical Faculty. Each patient will sign an informed consent prior to the inclusion into the prospective observational study.

In all patients, the thickness of the sternocleidomastoid muscle (SCM), trapezius muscle (TM), and quadriceps femoris (QF) muscle will be measured. A measurement point is in the middle of each muscle. The diameter of each muscle will be measured three times, and the average of the three measurements will be calculated.

In each patient hours of mechanical ventilation, and total time in the ICU will be recorded. Patients' comorbidities, ie. hypertension, cardiac diseases, diabetes, and other metabolic disorders, history of stroke, disabilities, as well as procedures done will be registered.

A Pearson's or Spearman's correlation will be used to calculate connections between specific parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with and without chronic respiratory diseases
* Mechanically ventilated patients
* Patients who gave consent to participate in the study

Exclusion Criteria:

* Patients with severe head and neck trauma
* Patients who have had upper leg surgery
* Patients who did not consent to participate in the study

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study was conducted on 50 patients admitted into the ICU. Patients of both genders were included, with and without chronic respiratory diseases, including mechanically ventilated patients.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Number of days in the ICU | Three months
  In order to be able to determine the outcome of treatment of patients in the intensive care unit, it is necessary to have a variable on how long the patients have been in the intensive care unit. Days spent in the ICU until discharge or death will be recorded.
Hours of mechanical ventilation | Three months
  Total hours spent on the mechanical ventilation is an important variable to compare with the treatment outcome of patients in the intensive care unit.
  Hours on mechanical ventilation until extubation will be recorded.
Accessory respiratory musculature thickness in patients with chronic lung disease and without chronic lung disease will be compared. | Three months
  An average of three measurements of accessory respiratory muscles, i.e. sternocleidomastoid (SCM) and trapezius muscle (TM) will be recorded.
  In addition, four heads of quadriceps femoris (QF) muscle will be measured three times and average of measurements will be recorded. A sum of all four heads will be registered in every patient. QF is usually a measure of patients' nutritive status and his/her mobility. It is expected to be thinner in the malnourished patients, in patients with mobility disorders and in older patients.
  A ratio between SCM, TM, and QF will be calculated for all the patients.
Relationship between quadriceps muscle (QM) thickness and patient age | Three months
  A correlation between patients' age and QM will be calculated.
Outcomes of the patients' treatment in the intensive care unit, will be recorded and correlated with QF, accessory respiratory muscles (SCM and TM) thicknes. | Three months
  A ratio between SCM and TM will be correlated with duration of the mechanical ventilation and total days in the ICU.

SECONDARY OUTCOMES:
An influence of patients' demographic characteristics will be recorded and correlated with muscle thickness and outcomes. | Three months
  For each patient age, sex, BMI, and comorbidities will be recorded, and correlated with hours of mechanical ventilation, days of ICU stay, and with accessory respiratory muscle thickness. A Pearson's or Spearman's correlation will be used for corelation analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Lea Atlagic, M.D., Principal Investigator — Osijek University Hospital; Medical Faculty
Locations (1):
- Osijek University Hospital, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: Yes
Once the study is completed the data will be publicly available.
Supporting Information: Study Protocol, CSR
Time Frame: once the study is published the data will be uploaded and permanently available and stored at ClinicalTrials.gov.
Access Criteria: public

REFERENCES:
- [Background] Pardo E, El Behi H, Boizeau P, Verdonk F, Alberti C, Lescot T. Reliability of ultrasound measurements of quadriceps muscle thickness in critically ill patients. BMC Anesthesiol. 2018 Dec 27;18(1):205. doi: 10.1186/s12871-018-0647-9. PMID 30591032
- [Background] Zhi H, Guo J, Zhao Y, Nie S, Li S, Wang S, Li Y. [Diagnostic accuracy of bedside ultrasound measurement of limb skeletal muscle thickness for intensive care unit-acquired weakness]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2020 Apr;32(4):494-497. doi: 10.3760/cma.j.cn121430-20200403-00084. Chinese. PMID 32527360
- [Background] Weijs PJ, Looijaard WG, Dekker IM, Stapel SN, Girbes AR, Oudemans-van Straaten HM, Beishuizen A. Low skeletal muscle area is a risk factor for mortality in mechanically ventilated critically ill patients. Crit Care. 2014 Jan 13;18(2):R12. doi: 10.1186/cc13189. PMID 24410863
- [Background] Gruther W, Benesch T, Zorn C, Paternostro-Sluga T, Quittan M, Fialka-Moser V, Spiss C, Kainberger F, Crevenna R. Muscle wasting in intensive care patients: ultrasound observation of the M. quadriceps femoris muscle layer. J Rehabil Med. 2008 Mar;40(3):185-9. doi: 10.2340/16501977-0139. PMID 18292919
- [Background] Nijholt W, Beek LT, Hobbelen JSM, van der Vaart H, Wempe JB, van der Schans CP, Jager-Wittenaar H. The added value of ultrasound muscle measurements in patients with COPD: An exploratory study. Clin Nutr ESPEN. 2019 Apr;30:152-158. doi: 10.1016/j.clnesp.2019.01.001. Epub 2019 Jan 29. PMID 30904216